CLINICAL TRIAL: NCT01339663
Title: Phase I Study To Evaluate The Use Of Autologous T- Antigen-Presenting Cells (T-APC) To Enhance The Persistence Of Adoptively Transferred CD8+ Antigen-Specific T Cells (CTL) Following Cyclophosphamide Conditioning For Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy Following Therapeutic Autologous Lymphocytes and Cyclophosphamide in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2481.00; NCI-2011-00383 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K12CA076930 (NIH)
Record Dates: First submitted 2011-04-18; First posted 2011-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; aldesleukin; Interleukin-2; FANG vaccine; Immunologic Techniques; Immunohistochemistry; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dose-escalation, T-APC boost, CTL) (Experimental): INFUSION I: Patients receive high-dose cyclophosphamide IV on day days -4 and -3 and low-dose IL-2 SC BID on days 0-14. Patients also receive CTL IV on day 0.
  INFUSION II: Beginning 6-48 hours later, patients receive high-dose cyclophosphamide, low-dose IL-2, and CTL as in Infusion I. Patients also receive T-APC vaccine IV within 18-36 hours following CTL infusion and in week 4, and IL-2 SC BID on days 0-14 following second T-APC vaccination.
  Interventions: Drug: cyclophosphamide; Biological: aldesleukin; Biological: autologous tumor cell vaccine; Other: laboratory biomarker analysis; Other: immunologic technique; Other: immunohistochemistry staining method; Genetic: polymerase chain reaction; Biological: therapeutic autologous lymphocytes

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: autologous tumor cell vaccine — Receive T-APC via IV
  Other Names: AC vaccine; ATCV; Autologous Cell Vaccine
Other: laboratory biomarker analysis — Correlative studies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Biological: therapeutic autologous lymphocytes — Receive adoptively transferred CD8+ antigen-specific T cell clones via IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells

SUMMARY:
This phase I trial studies the side effects and best dose of autologous T-antigen-presenting cells (T-APC) vaccine following therapeutic autologous lymphocytes (CTL) and cyclophosphamide in treating patients with metastatic melanoma. Aldesleukin may stimulate lymphocytes, such as CTL, to kill melanoma cells. Treating lymphocytes with aldesleukin in the laboratory may help the lymphocytes kill more tumor cells when they are put back in the body. Vaccines made from melanoma antigen may help the body build an effective immune response to kill tumor cells and may boost the effect of the CTL. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving T-APC vaccine after CTL and cyclophosphamide may be an effective treatment for melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and toxicity of T-APC vaccination following adoptive T cell therapy.

II. Evaluate the functional and numeric in vivo persistence of adoptively transferred cytotoxic t lymphocytes (CTL) followed by T-APC vaccination.

SECONDARY OBJECTIVES:

I. Evaluate the antitumor effect of adoptive T cell therapy followed by T-APC vaccination.

OUTLINE : This is a dose-escalation study of T-APC vaccine.

INFUSION I: Patients receive high-dose cyclophosphamide intravenously (IV) on days -4 and -3 and low-dose aldesleukin (IL-2) subcutaneously (SC) twice daily (BID) on days 0-14. Patients also receive CTL IV on day 0.

INFUSION II: Beginning 6-48 hours later, patients receive high-dose cyclophosphamide, low-dose IL-2, and CTL as in Infusion I. Patients also receive T-APC vaccine IV within 18-36 hours following CTL infusion and in week 4, and IL-2 SC BID on days 0-14 following second T-APC vaccination.

After completion of study treatment, patients are followed up for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological documentation of melanoma concurrent with the diagnosis of metastatic disease
* Tumor expression of melanocyte differentiation antigen (MDA: MART-1 = 2+ staining or > 25%) by immunohistochemistry (IHC)
* Expression of human leukocyte antigen (HLA)-A201
* Zubrod performance status of '0-1' at the time of treatment
* Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray, computed tomography [CT] scan)
* Normal cardiac stress test will be required for all patients with any history of cardiac disease

Exclusion Criteria:

* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to entry
* Serum creatinine > 1.6 mg/dL or Creatinine clearance < 75 ml/min
* Serum glutamic oxaloacetic transaminase (SGOT) > 150 IU or > 3x upper limit of normal
* Bilirubin > 1.6 mg/dL
* Prothrombin time > 1.5 x control
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in one second (FEV1) < 2.0 L or carbon monoxide diffusing capacity (DLco) (corr for hemoglobin [Hgb]) < 75% will be excluded
* Congestive heart failure
* Clinically significant hypotension
* Symptoms of coronary artery disease
* Presence of cardiac arrhythmias on electrocardiograph (EKG) requiring drug therapy
* Ejection fraction < 50 % (echocardiogram or multi gated acquisition scan [MUGA])
* Symptomatic central nervous system metastases greater than 1 cm at time of therapy; patients with 1-2 asymptomatic, less than 1 cm brain/central nervous system (CNS) metastases without significant edema may be considered for treatment
* Patients with active infections or oral temperature > 38.2 C within 72 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy
* Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 3 weeks prior to T cell therapy; (patients with bulky disease may undergo cytoreductive chemotherapy but treatment will be discontinued at least 3 weeks prior to T cell therapy)
* Clinically significant autoimmune disorders or conditions of immunosuppression; patients with acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV)-1 associated complex or known to HIV antibody seropositive or known to be recently polymerase chain reaction (PCR)+ for hepatitis are not eligible for this study; virology testing will be done within 6 months of T cell infusion; the severely depressed immune system found in these infected patients and the possibility of premature death would compromise study objectives
* Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 3 weeks prior to T cell therapy
* Current treatment with steroids
* Patients must not be receiving any other experimental drugs within 3 weeks of the initiation of the protocol and must have recovered from all side effects of such therapy
* Patients for whom we are unable to generate MART-1 specific T cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Treatment-related dose limiting toxicity (DLT) as defined by Grade 3 or greater unexpected toxicity by the NCI Common Toxicity Criteria (CTC) v4.0 | Up to 8 weeks after the T cell infusion
  Assessed at the maximum tolerated dose (MTD) or dose level immediately below the dose level for which the incidence of DLT was less than 35%.
In vivo persistence of adoptively transferred T cells | At 4 weeks
  Assessed by intrapatient comparison between the first (without T-APC) and second (with T-APC) CTL infusion. Descriptive statistics will be applied and t-tests of intrapatient in vivo T cell persistence between the two Infusions will be determined.

SECONDARY OUTCOMES:
Clinical response | Up to 8 weeks after second dose

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States